CLINICAL TRIAL: NCT02563301
Title: A Randomised Crossover Trial Comparing the McGrath Series 5 Videolaryngoscope With the Macintosh Laryngoscope in Patients With Cervical Spine Immobilisation
Brief Title: Videolaryngoscopy in Patients With Cervical Spine Immobilisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Lynsey Foulds, Specialty Registrar Anaesthetics, NHS Tayside
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2008AN01
Record Dates: First submitted 2015-09-25; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Intubation; Difficult
MeSH Terms: interventions — Laryngoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- McGrath Series 5 (Active Comparator): Videolaryngoscope used to perform indirect (video) laryngoscopy and tracheal intubation
  Interventions: Device: Laryngoscopy
- Macintosh (Active Comparator): Laryngoscope used to perform direct laryngoscopy and tracheal intubation
  Interventions: Device: Laryngoscopy

INTERVENTIONS:
Device: Laryngoscopy — After establishing full monitoring, inducing general anaesthesia and ensuring paralysis, laryngoscopy is performed and the patient's trachea is intubated.

SUMMARY:
Tracheal intubation is more difficult in patients in whom cervical spine immobilisation is maintained during tracheal intubation. The McGrath Series 5 videolaryngoscope offers a potential solution. The relatively short radius of the blade curvature combined with the internal arrangement of optimal components means that the glottis can be seen without the need for alignment of the oral, pharyngeal and tracheal axes.

The investigators propose that the McGrath Series 5 videolaryngoscope will improve the view of the larynx in patients with limited neck movements, making intubation quicker, easier and possibly safer.

ELIGIBILITY:
Inclusion Criteria:

* Elective procedure requiring tracheal intubation
* Over 16 years of age

Exclusion Criteria:

* Emergency procedure
* Less than 16 years of age
* Unable to consent
* Symptomatic gastro-oesophageal reflux disease
* Evidence of raised intracranial pressure
* Known pharyngeal pathology

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Cormack and Lehane laryngoscopy grade | 5 minutes

SECONDARY OUTCOMES:
Time to intubation | 5 minutes
Rate of successful tracheal intubation | 5 minutes
Incidence of complications | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lynsey T Foulds, MBChB, Principal Investigator — NHS Tayside
Locations (1):
- NHS Tayside, Tayside, United Kingdom